CLINICAL TRIAL: NCT03494309
Title: Comparison of Open Reduction With Internal Fixation and Closed Reduction With External Fixation of Mandibular Sub-Condylar Fractures
Brief Title: Open Versus Closed Reduction of Mandibular Sub-Condylar Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Samira S Baloch, Assistant Professor of Oral & Maxillofacial Surgery, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107/RC/KEMU
Record Dates: First submitted 2018-03-24; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Mandibular Fractures
Keywords: Mandibular Subcondylar Fractures; Mouth Opening; Open Reduction and Internal Fixation; Closed Reduction with External Fixation
MeSH Terms: conditions — Mandibular Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORIF (Experimental): Open Reduction & Internal Fixation
  Interventions: Procedure: Open Reduction & Internal Fixation
- CREF (Active Comparator): Closed Reduction & External Fixation
  Interventions: Procedure: Closed Reduction & External Fixation

INTERVENTIONS:
Procedure: Open Reduction & Internal Fixation — Patients underwent surgery and the fractures were reduced under direct vision followed by internal fixation with titanium plates and screws
  Arms: ORIF
Procedure: Closed Reduction & External Fixation — Patients underwent closed reduction of the fracture and external fixation by arch bars & guided elastics
  Arms: CREF

SUMMARY:
Patients with mandibular sub-condylar fractures underwent either either open reduction with internal fixation (ORIF) or closed reduction with external fixation (CREF) and were followed up for 6 months to assess treatment adequacy with the hypothesis that ORIF is superior to CREF.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-60 years
* Displaced Mandibular Subcondylar Fractures(MCFs) irrespective of multiple mandibular fractures.

Exclusion Criteria:

* Bilateral MCFs
* MCF with mid-facial fractures
* Insufficient bilateral dentition
* Medically unfit for surgery
* Old healed mandibular fractures
* History of previous mandibular surgery for the same indication

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-11-15 (Actual); Study Completion 2015-11-15 (Actual)

PRIMARY OUTCOMES:
Mouth Opening | 6 months
  Mouth Opening shall be determined by measuring the maximal distance between the edges of upper and lower incisors with fully opened mouth; the measurement shall be made in millimeters (mm) using vernier caliper and mouth opening of 35 mm or more shall be classified as "adequate"
Occlusion | 6 months
  Occlusion shall be determined by maximum "inter-cuspation" as observed by the surgeon and patient self-reporting and will be classified as fine or deranged.

SECONDARY OUTCOMES:
Complications | 6 months
  The frequency of complications with either mode of treatment shall be recorded
Cost-Effectiveness | 6 months
  Cost-Effectiveness shall be determined as the ratio of the cost of treatment and achievement of both adequate mouth opening and fine occlusion.
  The cost of treatment shall include the cost of surgical items (wires, elastics, arch bars, plates, screws etc), cost of anesthesia and surgery, cost of hospital stay and cost of follow up.
Patient Satisfaction | 6 months
  Participants shall be requested to report their satisfaction after treatment with regards to ease of chewing, mouth opening & closing and achievement of pre0traumatic facial symmetry/orientation.
  This parameter shall be recorded on a 4-point Likert scale (not satisfied, somewhat dissatisfied, somewhat satisfied, satisfied).